CLINICAL TRIAL: NCT07084935
Title: Comparison of the Surgical Pleth Index and the Nociception Level Index in the Pediatric Population: An Observational Study
Brief Title: Comparison of the Surgical Pleth Index and the Nociception Level Index in the Pediatric Population
Acronym: NOLvsSPI
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Ignacio Malagon, prof. Jose Ignacio Malagon Calle MD, PhD, Radboud University Medical Center
Other Study IDs: 2025-18010
Record Dates: First submitted 2025-07-02; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Nociceptive Pain; Anesthesia; Pediatric Anesthesia; Nociception Monitoring
Keywords: Nociception monitoring; Pediatric population; NOL index; Surgical pleth index
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 1 to 12 years undergoing surgery with general anesthesia.
  Interventions: Device: Connecting all patients to the nociception level index(NOL) and the surgical pleth index (SPI); Device: All patient will receive a tetanic stimuli (60mA, 100hz) of 5 seconds before start of incision

INTERVENTIONS:
Device: Connecting all patients to the nociception level index(NOL) and the surgical pleth index (SPI) — All patients will be connected to the NOL and SPI during surgery after induction of general anesthesia.
Device: All patient will receive a tetanic stimuli (60mA, 100hz) of 5 seconds before start of incision — All patient will receive a tetanic stimuli (60mA, 100hz) of 5 seconds before start of incision.

SUMMARY:
This observational study aims to compare two nociception monitoring methods. The Nociception Level (NOL) index and the Surgical Pleth Index (SPI) in the pediatric population during general anesthesia. While both monitors are designed to assess nociceptive responses through autonomic nervous system activity, they differ in methodology and parameters measured. The NOL index integrates multiple physiological signals using a self-learning algorithm, while SPI focuses on heart rate variability and plethysmographic amplitude. Although both have been studied individually in children, a direct comparison has not yet been conducted. This study will evaluate and compare each monitor's ability to detect and quantify nociceptive stimuli (surgical and tetanic) in children.

The investigators hypothesize that the NOL monitor and SPI monitor will both be able to quantify surgical stimuli and tetanic stimuli with monitors response to surgical stimuli > monitors response to tetanic stimuli. However, the investigators also hypothesize that the NOL index will do this superiorly, as it utilizes a self-learning algorithm and more parameters are incorporated in its algorithm

DETAILED DESCRIPTION:
This is a single centre, observational prospective non-interventional study. The study will take place at the Radboudumc. After obtaining informed consent participants will be enrolled. Each participant will be treated according to the standard Radboudumc anaesthesia protocol with heartrate monitoring, respiratory rate monitoring, neuromuscular monitoring (TOF-Watch SX ) , intermittent non-invasive blood pressure monitoring and Bispectral index monitoring. Participants will be connected to the NOL index PMD-200 device using the finger probe and the SPI device (Carescape b650) using the pulse oxymeter directly after induction of anesthesia with propofol/sevoflurane. Before start of surgery, after recording a period of 30 seconds with no stimulation (no nociception) a standardised tetanic stimulus of 5 seconds with 60 mA and 100hz will be applied with the neuromuscular monitor on the patients ulnary nerve trajectory with two adhesive electrodes. This is a stimulus that is part of common anesthesiology practice in order to assess the patients neuromuscular blockade. Previous research has used tetanic stimuli of similar intensity as standardised nociceptive stimuli in order to validate nociception monitors. After SPI and NOL monitor values return to baseline (pre-tetanic stimulus value) surgery with first incision will commence.

During the operation the response to the standardised stimuli and nociceptive events such as intubation, insertion of supraglottic airway, surgical incision and administration of opioids will be registered by a trained researcher. After surgery, upon discharge to the anaesthesia recovery room, patients will be disconnected from both monitors. Post-operative pain/comfort scores and post-operative analgesia usage will be registered by the researcher at the recovery room. Total duration of the study inclusion period is expected to be 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ASA I, ASA II and ASA III
* Aged 1 to 12 years old
* Scheduled to undergo elective surgery with general anaesthesia

Exclusion Criteria:

* Patients with chronic pain
* Patients with chronic analgesia usage.
* Known allergy to the adhesives used in the sensors.
* No free available limb to attach the probes to.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients scheduled to undergo surgery with general anesthesia at the Radboud university medical centre in Nijmegen, the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in surgical pleth index (∆SPI) during surgical stimuli and standardized tetanic stimuli | During surgery with general anesthesia.
  ∆SPI = pre stimulus -30s-0s mean SPI value - post stimulus +5s to 30s-120s SPI value.
Change in nociception level index (∆NOL) during surgical stimuli and standardized tetanic stimuli | During surgery with general anesthesia
  ∆NOL = pre stimulus -30s-0s mean NOL value - post stimulus +5s to 30s-120s NOL value.

SECONDARY OUTCOMES:
Change in surgical pleth index (∆SPI) following intraoperative opioid administration. | During surgery with general anesthesia]
  Response of the SPI to intraoperative administration of opioids. Evaluate SPI mean values -20s to 0s before opioid administration to mean value after opioid administration in accordance with the utilized opiod farmacokinetics(time of mean measurement in seconds depends on opioid used).
Change in nociception level index (∆NOL) following intraoperative opioid administration. | During surgery with general anesthesia
  Response of the NOL index to intraoperative administration of opioids. Evaluate NOL mean values -20s to 0s before opioid administration to mean value after opioid administration in accordance with the utilized opiod farmacokinetics(time of mean measurement in seconds depends on opioid used).
Time NOL index is >25 and SPI is >40 during surgery and before intra-operative opioid administration. Defined as time NOL index is >20-25 and SPI is >40 during surgery time. | During surgery with general anesthesia
  Defined as time in seconds NOL index is >25 and SPI is >40 during surgery time.
Comparing mean (total surgery time) and last 5-min mean values before disconnection for intra-operative NOL and SPI to the post-operative pain scores. | perioperative/periprocedural
  * For patients aged <4 Faces, legs, activity, cry and consolability (FLACC) will be used
  * For patients aged >4 a faces pain scale, numeric rating scale (NRS) or visual analogue scale (VAS) will be used.
  * Pain scores will be obtained at recovery admittance, after one hour and at recovery departure and when recovery personnel deem it is necessary based on their clinical view.
Change in surgical pleth index (∆SPI) after administration of vasoactive medication. | During surgery with general anesthesia
  Compare mean values -20 to 0 sec for administration of vasoactive medication to mean 5+-30 sec, 5+-60sec and 5+-120sec after administration vasoactive medication (noradrenaline, ephedrine and atropine).
Change in nociception level index (∆NOL) after administration of vasoactive medication. | During surgery with general anesthesia
  Compare mean values -20 to 0 sec for administration of vasoactive medication to mean 5+-30 sec, 5+-60sec and 5+-120sec after administration vasoactive medication (noradrenaline, ephedrine and atropine).
Change in heartrate (∆HR) following a nociceptive event and opioid administration. | During surgery with general anesthesia
  Change in heartrate following a nociceptive event. pre stimulus -30s-0s mean HR value - post stimulus +5s to 30s-120s HR value.
  Following opioid administration:
  Change in heartrate mean values -20s to 0s before opioid administration to mean value after opioid administration in accordance with the utilized opiod farmacokinetics(time of mean measurement in seconds depends on opioid used).
Change in mean arterial bloodpressure(∆MAP) following nociceptive event and opioid administration | During surgery with general anesthesia
  Comparision of mean arterial bloodpressure measurement before nociceptive event/opioid administration to measurement after nociceptive event/opioid administration.
Change in respiratory rate (∆RR) following a nociceptive event and opioid administration. | During surgery with general anesthesia
  Change in respiratory rate following a nociceptive event. pre stimulus -30s-0s mean HR value - post stimulus +5s to 30s-120s HR value.
  Following opioid administration:
  Change in respiratory rate mean values -20s to 0s before opioid administration to mean value after opioid administration in accordance with the utilized opiod farmacokinetics(time of mean measurement in seconds depends on opioid used).
Change in nociception level index (Δ NOL) after incision under loco-regional/neuraxial blockade. | During surgery with general anesthesia.
  Defined as Δ NOL following nociceptive stimuli in patients with an active loco-regional or neuraxial blockade.
  Compare mean values of SPI and NOL -30-0 before incision to mean 5+-30 sec, 5+-60sec and 5+-120sec after incision.
Change in surgical pleth index (Δ SPI) after incision under locoregional/neuraxial blockade. | Δ SPI
  Defined as Δ SPI following nociceptive stimuli in patients with an active loco-regional or neuraxial blockade.
  Compare mean values of SPI and NOL -30-0 before incision to mean 5+-30 sec, 5+-60sec and 5+-120sec after incision.
Response time of both monitors after nociceptive stimulation. | During surgery with general anesthesia
  Defined as time in seconds of onset to change in SPI and NOL after nociceptive stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Malagon, Professor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided